CLINICAL TRIAL: NCT05208450
Title: Actions to Decrease Disparities in Risk and Engage in Shared Support for Blood Pressure Control (ADDRESS-BP) in Blacks
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20-01114
Record Dates: First submitted 2022-01-11; First posted 2022-01-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-06

CONDITIONS: Hypertension (HTN)
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (UC) Group (No Intervention): The study design is a randomized stepped wedge cluster trial whereby all clusters (practice sites) begin as part of the Usual Care (UC) control condition.
  Clusters are then randomly assigned to cross over at different times with all clusters eventually receiving PACE. The study will involve each site starting with the UC, followed by a period of 3 months during which practice facilitators will train NCMs and CHWs, and finally followed by the PACE intervention for 12 months with a 6-month follow-up for outcome assessment. During the UC Period, patients at the sites will receive standard HTN care and standard printed HTN treatment guidelines. Immediately following this period, prior to implementation of PACE, we will conduct a practice capacity assessment at each site for 3 months. This period is then followed by the implementation of PACE.
- Intervention Group (Experimental): Thus, each cluster will belong successively to the control group and the intervention group. During the control period (UC) patients at the sites will receive standard HTN care delivered by their primary care providers and standard printed HTN treatment guidelines. This period is then followed by the implementation of PACE. Clusters are randomly assigned to cross over at different times with all clusters eventually receiving PACE. During the PACE implementation period, which will last 12 months, practice facilitators will work with each site to implement the components of PACE.
  Interventions: Other: Practice support And Community Engagement (PACE)

INTERVENTIONS:
Other: Practice support And Community Engagement (PACE) — A practical and sustainable implementation strategy, referred to as Practice Facilitation And social deTerminants of health support utilizing CHWs (PATCH), to support the implementation and evaluation of three multi-level evidence-based interventions: [nurse case management (NCM) + remote blood pressure monitoring (RBPM) + social determinants of health (SDOH) support] delivered as an integrated community-clinic linkage model [Practice support And Community Engagement (PACE)]
  Arms: Intervention Group

SUMMARY:
To use practice facilitation (PF) + community health worker (CHW) facilitation as a practical and sustainable implementation strategy to support the implementation and evaluation of three multi-level evidence-based interventions [nurse case management (NCM), remote blood pressure monitoring (RBPM), and social determinants of health (SDOH) support] delivered as an integrated community-clinic linkage model [Practice support And Community Engagement (PACE) to address patient-, physician-, health system-, and community-level barriers to hypertension (HTN) control in Blacks across 25 primary practices within NYU Langone Health in New York City (NYC) and, in partnership with an established Community-Clinic-Academic Advisory Board and HealthFirst (NYC's largest Medicaid payer).

The goal for the UH3 Implementation Phase (Years 4-7, Intervention) is to evaluate a stepped-wedge cluster RCT of 25 primary care practices in Black patients with uncontrolled hypertension (HTN)

ELIGIBILITY:
UH3 IMPLEMENTATION PHASE (Years 4 - 7): INTERVENTION

Inclusion Criteria:

Patients are eligible if he/she:

1. identifies as Black (through EHR code or self-report)
2. is 18+ years of age
3. has a diagnosis of HTN (identified by ICD-10 codes for HTN)
4. prescribed an antihypertensive medication(s)
5. has a clinic BP > 130/80 mmHg

Exclusion Criteria:

Patients will be ineligible for the study if they:

1. are deemed unable to comply with the study protocol (either self-selected or by indicating during screening that s/he could not complete all requested tasks)
2. participate in other hypertension-related clinical trials
3. have significant psychiatric comorbidity or reports of substance abuse (as documented in the EHR)
4. plan to discontinue care at the site within the next 12 months; or
5. are pregnant or planning to become pregnant in the next 12 months

IMPLEMENTATION EVALUATION

1. NYULH Primary care provider (MD/DO, NP), Clinical Director, Site Administrator, Medical Assistant, or administrative staff employed at the participating practices and interacts with at least five patients with a diagnosis of hypertension; or
2. NYULH Nurse case manager within centralized service; or
3. Staff and leadership of community- and faith-based organizations serving the Black community; or
4. NYULH Organizational leadership; or
5. NYULH Project Staff: Community Health Workers/CHW Supervisor/Practice Facilitators; and
6. Able and willing to provide consent

Exclusion Criteria:

1. Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of Nurses who adopt the PACE intervention | Month 12
  Defined at the Nurse-level who adopt both electronic health record (EHR) remote BP monitoring (RBPM) and social determinants of health (SDOH) Smartsets

CONTACTS AND LOCATIONS:
Overall Officials: Gbenga Ogedegbe, MD, MPH, Principal Investigator — NYU Langone Health; Nadia Islam, PhD, Principal Investigator — NYU Langone Health; Antoinette Schoenthaler, EdD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to data upon reasonable request. Requests should be directed to Jennifer.zanowiak@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Gyamfi J, Cooper C, Barber A, Onakomaiya D, Lee WY, Zanowiak J, Mansu M, Diaz L, Thompson L, Abrams R, Schoenthaler A, Islam N, Ogedegbe G. Needs assessment and planning for a clinic-community-based implementation program for hypertension control among blacks in New York City: a protocol paper. Implement Sci Commun. 2022 Sep 6;3(1):96. doi: 10.1186/s43058-022-00340-z. PMID 36068611